CLINICAL TRIAL: NCT00571181
Title: Target-Controlled Infusion of Propofol and Remifentanil During General Anaesthesia Guided by the Index Bispectral: Comparison Between Manual Perfusion and Automated Perfusion During Rigid Bronchoscopy
Brief Title: Automated Anesthesia During Bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/14; EudraCT 2007-003157-82
Record Dates: First submitted 2007-12-09; First posted 2007-12-11 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia, General
Keywords: Algorithms; Anesthesia, General/*methods; Anesthetics, Intravenous/*administration & dosage; Drug Delivery Systems/*methods/statistics & numerical data; Electroencephalography/drug effects/*methods/; Feasibility Studies; Propofol/*administration & dosage; Remifentanil/*administration & dosage; Bronchoscopy/*methods; Prospective Studies; Software

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Closed-loop system
- 2 (Active Comparator)
  Interventions: Device: TCI (Infusion Toolbox)

INTERVENTIONS:
Device: Closed-loop system — Automatic delivery of propofol and remifentanil
  Arms: 1
Device: TCI (Infusion Toolbox) — TCI administration of propofol and remifentanil
  Arms: 2

SUMMARY:
The purpose of this study is to compare manual administration of propofol and remifentanil and dual closed-loop using bispectral index as the control variable during rigid bronchoscopy.

DETAILED DESCRIPTION:
The Bispectral Index (BIS) is an electroencephalogram-derived measure of anesthetic depth. We have built a combined closed-loop anesthesia system using BIS as the control variable, two proportional-integral-differential control algorithms, a propofol and a remifentanil target-controlled infusion systems as the control actuators. A recent study has shown that such system is able to provide clinically adequate anesthesia. The aim of the present study is to assess the system during rigid bronchoscopy. Two groups of patients are compared: one in which propofol and remifentanil are administered by the anesthesiologist using target-controlled infusion systems, and one in which propofol and remifentanil are administered automatically by the combined closed-loop anesthesia system. In both groups, the goal is to maintain BIS between 40 and 60, the recommended range during anesthesia by the manufacturer. We expect the combined closed-loop anesthesia system group to do similar or better.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing rigid bronchoscopy under general anesthesia

Exclusion Criteria:

* pregnant women
* allergy to propofol or remifentanil
* neurological disorder
* psychotrop treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Percentage of time with BIS in the desired range | During the procedure

SECONDARY OUTCOMES:
consumption of propofol and remifentanil | during the procedure
extubation time | during the procedure
explicit memorisation | postoperative day 2

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (1):
- Service d'Anesthésie, Hôpital Foch, Suresnes, France

REFERENCES:
- [Background] Liu N, Chazot T, Trillat B, Pirracchio R, Law-Koune JD, Barvais L, Fischler M. Feasibility of closed-loop titration of propofol guided by the Bispectral Index for general anaesthesia induction: a prospective randomized study. Eur J Anaesthesiol. 2006 Jun;23(6):465-9. doi: 10.1017/S0265021506000196. PMID 16672092
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Derived] Liu N, Pruszkowski O, Leroy JE, Chazot T, Trillat B, Colchen A, Gonin F, Fischler M. Automatic administration of propofol and remifentanil guided by the bispectral index during rigid bronchoscopic procedures: a randomized trial. Can J Anaesth. 2013 Sep;60(9):881-7. doi: 10.1007/s12630-013-9986-7. Epub 2013 Jul 16. PMID 23857041